CLINICAL TRIAL: NCT01432860
Title: A Comparison of Interventions to Teach Melanoma Patients Skin Self-examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STU17005
Record Dates: First submitted 2011-08-15; First posted 2011-09-13 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma
Keywords: Skin Self Examination
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- In-person Counseling and Education (Active Comparator): In the in-person training the Research Assistant demonstrates the use of a mm ruler, a lighted magnifying lens, a set of body maps and a scorecard, 4 pens, ABCDE rule on the skin exam card and discusses the ABCDE rule by pointing to the color examples on the skin exam card. 165 pairs (330 subjects) are randomized to this arm.
  Interventions: Behavioral: In-person counseling
- Workbook (Active Comparator): The workbook, which includes all of the information delivered in the in-person intervention, is 39 pages in length, and has 76 color figures. Each element of the in-person training represents a chapter in the workbook. The introduction explores the partners' understanding of melanoma and their personal risk of developing another melanoma, and attitudes about the benefit of early detection assisted by a partner. The early detection segment uses a skin diagram to illustrate the difference between thin and thick melanoma and presents the treatment based on the depth of the melanoma. 165 pairs (330 subjects) are randomized to this arm.
  Interventions: Behavioral: Workbook
- Control (No Intervention): Education and counseling as usually delivered in clinical practice. 100 pairs (200 subjects) are randomized to this arm.
- Tablet Computer-Based Education (Active Comparator): Education will be given by an interactive tablet app. Each pair will view video recordings of certain parts of the in-person presentation as well as select slides from the in-person PowerPoint presentation. Parts of the workbook will be incorporated as well. 70 pairs (140 subjects) are randomized into this arm.
  Interventions: Behavioral: Tablet Computer-Based Education

INTERVENTIONS:
Behavioral: In-person counseling — The design is a 3 [in-person training of patients and partners (PARTNER) vs. workbook training of patients and partners (WORKBOOK) vs. an assessment only group that receives education and treatment as usual care] X 7 [baseline, 4, 8, 12, 16, 20, and 24 month follow-up] study. Standard education of melanoma patients, which are to be performed with the study partner, includes a recommendation to check moles and mark ones to remember on a body map. All participants receive the same measures and will be recruited using the same procedures, thus, yielding equivalence across conditions. Pairs will observe how to use their skin check tools and be asked to demonstrate their competence in using them.
  Arms: In-person Counseling and Education
Behavioral: Workbook — Participants will read a workbook and perform skills training exercises.
  Arms: Workbook
Behavioral: Tablet Computer-Based Education — Participants will receive their education from an interactive app designed for a tablet computer.
  Arms: Tablet Computer-Based Education

SUMMARY:
The almost 724,000 Americans survivors of melanoma are estimated to have 4 first degree relatives per case; thus, 2.8 million Americans are at increased risk of developing melanoma in comparison to the general public. Skin self-examination (SSE) with the assistance of a partner by these individuals could improve survival. If effective, the workbook tested in this proposal could be distributed to people at risk of developing melanoma by large scale means in physicians office.

DETAILED DESCRIPTION:
Population based registries document that survival from melanoma, a growing public health problem with approximately 70,000 new melanoma cases and an estimated 8,600 deaths in 2010, is dependent on the thickness of the melanoma. By facilitating seeking medical care, skin self-examinations (SSEs) by individuals with a prior history of melanoma, who are at risk to develop subsequent melanomas, may lead to the early detection and treatment of melanoma when it is usually more effective. Thus, further research that enhances early detection is warranted and our application directly tests novel methods of training high-risk melanoma patients and their partners on how to conduct SSEs to promote early detection. Our proposed research builds upon the strengths of the R21 that: a) established that in-person training to conduct SSE with a partner significantly enhanced SSE performance 4 months after the intervention, and b) developed and pilot tested a manualized take-home workbook training approach (WORKBOOK). Our pilot work on the WORKBOOK with partners suggests that patient-partner dyads (n = 21) perceived it to be readable, useful, and in the short term 4 month follow-up, empirically equivalent in promoting SSE knowledge, skills, and behaviors compared with patient-partner dyads in the in-person partner training condition (n = 19). Our proposed research builds on our NCI funded studies by conducting a formal examination with 430 pairs (860 subjects) randomized to either the in-person or workbook training vs. an assessment only control group that receives standard of care over a 2 year longitudinal study with 4 month interval evaluations. An additional group of 70 pairs (140 subjects) has been added to test a tablet computer-based program.

Our proposed research directly tests novel methods of training Stage I and IIB melanoma patients, who have a 5 year survival of 80-90%, and their partners, on how to conduct SSEs. We will compare the efficacy of the in-person training vs. workbook for patients and partners vs. controls on SSE knowledge/skill acquisition and retention, and SSE performance and accuracy on a short (4 and 8 months post baseline) and long term basis (12, 16, 20, and 24 months post baseline) and examine whether partner-patient relationship-qualities moderate the relationship between the training approaches and SSEs knowledge/skill acquisition and retention, and SSE performance and accuracy. The tablet computer-based program will also be tested for efficacy and compared with the previous groups.

Establishing health promotion partnerships is important to those at risk to develop melanoma because SSE is difficult to successfully perform as an individual. It is expected that the workbook will promote SSE at least as well as and perhaps better than in-person training and become an easily disseminated SSE training approach that is not dependent on the time and teaching skills of the non-MD clinical office staff.

ELIGIBILITY:
Inclusion Criteria:

1. Personal history of Stage 0 through IIB melanoma
2. At least 6 weeks post surgical treatment of Stage 0 through IIA melanoma
3. Age 18-80 years old
4. Have sufficient vision to read a newspaper in order to visually detect changes on skin
5. Able to read English
6. Have a partner willing to participate in skin checks

Exclusion Criteria:

1.Subjects overburdened with other co- morbid diseases, medical treatments (e.g. chemotherapy), unable to participate in a conversation at a sixth grade language level due to cognitive impairment (e.g. by a stroke), or prior participation in SSE research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy in Performing SSE | 24 months
  To compare the self-efficacy of the in-person training vs. workbook for patients and partners by self-report on a survey at 4-month intervals over 24 months.

SECONDARY OUTCOMES:
Accuracy | 24 months
  Accurate identification of concerning lesions (melanoma) by participants performing SSE in comparison with the dermatologist's assessment.

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
publication of results with listing in My NCBI

REFERENCES:
- [Background] Hultgren BA, Turrisi R, Mallett KA, Ackerman S, Robinson JK. Influence of Quality of Relationship Between Patient With Melanoma and Partner on Partner-Assisted Skin Examination Education: A Randomized Clinical Trial. JAMA Dermatol. 2016 Feb;152(2):184-90. doi: 10.1001/jamadermatol.2015.2819. PMID 26422745
- [Background] Robinson JK, Wayne JD, Martini MC, Hultgren BA, Mallett KA, Turrisi R. Early Detection of New Melanomas by Patients With Melanoma and Their Partners Using a Structured Skin Self-examination Skills Training Intervention: A Randomized Clinical Trial. JAMA Dermatol. 2016 Sep 1;152(9):979-85. doi: 10.1001/jamadermatol.2016.1985. PMID 27367303
- [Result] Stapleton JL, Turrisi R, Mallett KA, Robinson JK. Correspondence between pigmented lesions identified by melanoma patients trained to perform partner-assisted skin self-examination and dermatological examination. Cancer Epidemiol Biomarkers Prev. 2015 Aug;24(8):1247-53. doi: 10.1158/1055-9965.EPI-15-0218. Epub 2015 Jun 10. PMID 26063475
- [Result] Turrisi R, Hultgren B, Mallett KA, Martini M, Robinson JK. Comparison of Efficacy of Differing Partner-Assisted Skin Examination Interventions for Melanoma Patients: A Randomized Clinical Trial. JAMA Dermatol. 2015 Sep;151(9):945-51. doi: 10.1001/jamadermatol.2015.0690. PMID 26049533
- [Result] Rikki G, Brittney H, Jerod S, Mallett Kimberly A, Rob T, Claudia H, Karl B, Wayne Jeffrey D, Martini Mary C, Robinson June K. The Influence of Disease Perceptions on the Participation of Melanoma Patients and their Partners in Skin Self-Examination Education. J Community Med Health Educ. 2013 Nov 1;3(6):242. doi: 10.4172/2161-0711.1000242. PMID 24795843
- [Result] Gaber R, Mallett KA, Hultgren B, Turrisi R, Gilbertsen ML, Martini MC, Robinson JK. Enhanced fidelity of an educational intervention on skin self-examination through surveillance and standardization. J Nurs Educ Pract. 2014;4(2):253-258. doi: 10.5430/jnep.v4n2p253. PMID 25414761
- [Result] Robinson JK, Gaber R, Hultgren B, Eilers S, Blatt H, Stapleton J, Mallett K, Turrisi R, Duffecy J, Begale M, Martini M, Bilimoria K, Wayne J. Skin self-examination education for early detection of melanoma: a randomized controlled trial of Internet, workbook, and in-person interventions. J Med Internet Res. 2014 Jan 13;16(1):e7. doi: 10.2196/jmir.2883. PMID 24418949